CLINICAL TRIAL: NCT00959387
Title: Induction Chemotherapy (IC) With Paclitaxel and Cisplatin (PC) Followed by Concomitant Chemoradiotherapy (CCRT) in Patient With Advanced Squamous Carcinoma of the Head and Neck (SSCHN).
Brief Title: Induction Chemotherapy for Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Luciano de Souza Viana, MD, PhD, Barretos Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Barretos-01
Record Dates: First submitted 2009-08-03; First posted 2009-08-14 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; induction chemotherapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Paclitaxel; Cisplatin; Chemoradiotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Induction TP chemotherapy followed by CRT (Experimental): paclitaxel 175mg/m2 as a 3-h infusion on Day 1, and cisplatin 80mg/m2 as a 2-h infusion on Day 1 three weekly followed by concurrent chemoradiotherapy based on cisplatin. All patient were given adequate hydration and antiemetics. All patients received supportive care during radiotherapy, including dietary measures, local antiseptics and laser therapy as preventive and curative support for oral mucositis.
  Interventions: Drug: Induction TP chemotherapy; Radiation: Chemoradiotherapy (CRT)

INTERVENTIONS:
Drug: Induction TP chemotherapy — 3 cycles of paclitaxel 175mg/m2 and cisplatin 80mg/m2 q3w. All patients received supportive care during radiotherapy, including dietary measures, local antiseptics and laser therapy as preventive and curative support for oral mucositis.
  Other Names: Paclitaxel; Cisplatin
Radiation: Chemoradiotherapy (CRT) — Patients were treated with 2-dimensional radiation therapy planning (6MV photon beams). A combination of lateral-opposed portals, anterior and lateral wedged fields was used to treat the primary tumor and the lymph nodes. The primary tumor, macroscopically affected lymph nodes and bilateral cervical plus supraclavicular lymph chains were treated with five fractions of 2Gy per week for 5 weeks (up to a total of 50Gy). Gross tumor volume was defined as the primary gross tumor or involved node, and this measure was based on clinical, radiological and endoscopic examinations. An additional margin of 1.0cm was added to the GTV to create the CTV. A boost of five fractions of 2Gy per week for 2 additional weeks (up to a total dose of 70Gy) was prescribed to the CTV plus a margin of 1.0cm.
  Other Names: Cisplatin; Radiotherapy; Concurrent chemoradiotherapy based on cisplatin

SUMMARY:
Over the last 30 years, induction chemotherapy (IC) has become important for the management of patients with locally advanced HNSCC (LAHNSCC), particularly since the introduction of taxanes. The results reported in the TAX 323 and TAX 324 trials indicate that the TPF regimen (docetaxel, cisplatin and 5-fluorouracil) improves overall survival comparing with the PF regimen (cisplatin and 5-fluorouracil), and the TPF regimen is globally the most accepted induction regimen for the treatment of LAHNSCC.

However, the TPF regimen has been associated with high toxicity rates, and patients frequently decline cisplatin during concurrent radiotherapy and require the use of infusion pumps and a central venous catheter.

Extensive efforts are ongoing to identify alternative schemes that are less toxic than the TPF regimen but are as effective for LAHNSCC and safely allow the use of definitive concurrent treatment based on cisplatin and radiotherapy.

DETAILED DESCRIPTION:
This non-randomized phase II trial evaluated the safety, feasibility and response rates of concurrent therapy (cisplatin and radiotherapy) after three cycles of an IC regimen based on the combination of cisplatin plus paclitaxel without 5-fluorouracil (5FU) (thereby avoiding infusion pumps and a central venous catheter) in LAHNSCC patients with a high tumor burden.

The patients were stratified by tumor subsite (oropharynx and hypopharynx/larynx) and by tumor resectable status (resectable or irresectable advanced squamous cell).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed locally advanced squamous cell carcinoma of head and neck (stage III and IV) eligible to chemoradiotherapy.
* Presence of measurable disease
* ≥ 18 year
* ECOG performance status: 0-2
* Adequate bone marrow functions evidenced by: absolute neutrophil count ≥ 1.5 x 109/L; platelet count ≥ 100 x 109/L and hemoglobin ≥ 90 g/L
* Adequate renal function.
* Adequate hepatic function.
* Patients or their legal representatives must be able to read, understand and provide written informed consent to participate in the study.

Exclusion Criteria:

* Any previous chemotherapy or radiotherapy
* Patients who have known hypersensitivity to paclitaxel or cisplatin
* Patients who are receiving concurrent investigational, biological or immune therapies
* Concomitant administration of high doses of systemic corticosteroids
* Known HIV or Hepatitis B or C (active, previously treated or both; testing is not required)
* Uncontrolled CNS disease (e.g., seizures not controlled with standard medical therapy)
* Clinically significant cardiovascular disease.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-08; Primary Completion 2010-11 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Tumor response rate | At baseline, 2 weeks after the third cycle of IC and 6-8 weeks after the end of radiotherapy
  Tumor response was assessed after induction chemotherapy (just before chemoradiotherapy) and 6-8 weeks after completion of chemoradiotherapy.
  Evaluation of tumor response was by clinical examination, nasoendoscopy, and CT or MRI imaging of the primary site and the neck (RECIST criteria 1.1).

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival (OS) was calculated as the time of study entry to the date of death.
Quality of life (EORTC QLQ-C30) | 2 years
  Questionnaire of quality of life (EORTC QLQ-C30) was applied at baseline, before chemoradiotherapy and 60 days following last day of radiotherapy.
Adverse Events rate | After every cycle of IC, after every cycle of concurrent chemetherapy and up to 8 weeks after the end of radiotherapy
  Adverse events were graded according to the expanded common toxicity criteria of the Clinical Trials Group of the National Cancer Institute of Canada (NCI CTCAE v3.0). Laboratory safety data were assessed before the administration of chemotherapy and after treatment.
Progression-free survival. | 3 years
  Progression-free survival (PFS) was calculated as the date of assignment to recurrence/progression or death resulting from any cause. If the patient had no evidence of the aforementioned events, survival was censored at the time of the last documented evaluation of efficacy/contact or death resulting from another cause.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano S Viana, MD, MSc, PhD, Principal Investigator — Brazilian Society of Clinical Oncology
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil